CLINICAL TRIAL: NCT05744167
Title: Resistance Training and Muscle - Brain Crosstalk
Brief Title: Blood Flow Restriction and High-intense Resistance Training in Aging: Interactions Between Neuroplasticity and Muscle
Acronym: BRAIN-M
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lithuanian Sports University (Other)
Collaborators: Research Council of Lithuania (Other); Lithuanian University of Health Sciences (Other); Maastricht University (Other); Vrije Universiteit Brussel (Other); KU Leuven (Other); Wingate Institute (Other)
Responsible Party: Principal Investigator, Vilma Dudoniene, Associated professor, Lithuanian Sports University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LithuanianSportsU-11
Record Dates: First submitted 2022-09-08; First posted 2023-02-24 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-08

CONDITIONS: Aging; Cognitive Decline; Sarcopenia; Frailty; Muscle Degeneration; Physical Disability
Keywords: Aging; Motor control; Cognitive function; Neuroplasticity; Brain health; Muscular fitness; Exerkines; Myokines; (Neuro)inflammation
MeSH Terms: conditions — Cognitive Dysfunction; Sarcopenia; Frailty

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Blood flow restriction training (BFRT) (Experimental): Participants will engage in a supervised 12-week lower extremity resistance exercise program, 2 times per week. BFRT will be at an intensity of 40% of 1RM with an occlusive cuff placed at the proximal end of both lower extremities to restrict the return of blood flow. The cuff will be inflated to 50% of the limb occlusion pressure in the first week, which will be increased with 10% every week during the first 4 weeks to reach a maximum of 80% limb occlusion pressure on week 4 that will be kept for the remaining 9 weeks of the program. Each exercise will be performed for 4 sets of 12 repetitions with a 30-second rest period between sets and 3 minutes rest between exercises without occlusion.
  Interventions: Behavioral: BFRT
- Muscle damaging resistance training (MDRT) (Experimental): Participants will engage in a supervised 12-week lower extremity resistance exercise program, 2 times per week. MDRT will be at an intensity of 80% or 120% of 1RM. The first session will be at 120% 1RM and consist of eccentric-only exercises. The concentric phase of the movement will be supported completely by a coach. The eccentric phase of the movement will be accentuated by increasing the time under tension to six seconds. Each exercise will be performed for 4 sets of 4 repetitions with 2 minutes rest between sets and 3 minutes rest between exercises. The eccentric-only exercise session will be followed by 2 (after the first session) or 3 (after all other sessions) concentric-only exercise sessions at 80% of 1RM. Here, the eccentric phase of the movement will be supported completely by a coach. In the 12 week period, there will be a total of seven eccentric-only exercise sessions.
  Interventions: Behavioral: MDRT
- Control group (No Intervention): Control group will be asked to maintain their usual lifestyle.

INTERVENTIONS:
Behavioral: BFRT — Following a warm-up of 10 min, subjects in the experimental group will undergo BFRT for two times per week, consisting of lower extremity exercises (leg press, knee extension, knee flexion). BFRT will be at 40% of 1 repetition maximum (1RM); The volume % (V% = number of repetitions x number of sets x number of exercises x % 1 repetition max) = 57.6%. Progression during the 12 week program will be attained by a 1RM test every 4 weeks.
  Arms: Blood flow restriction training (BFRT)
Behavioral: MDRT — Following a warm-up of 10 min, subjects in the experimental group will undergo MDRT for two times per week, consisting of lower extremity exercises (leg press, knee extension, knee flexion). The exercise will be at 80% of 1RM concentric-only or 120% of 1RM eccentric-only in a 3:1 ratio. The volume % (V% = number of repetitions x number of sets x number of exercises x % 1 repetition max) = 57.6%. Progression during the 12 week program will be attained by a 1RM test every 4 weeks.
  Arms: Muscle damaging resistance training (MDRT)

SUMMARY:
BRAIN-M is a randomized controlled trial designed to examine the effects of a single bout or 12 weeks of blood-flow restriction training or high-intensity resistance training on cognitive function, brain health, muscular properties and physical performance in healthy older men 60-75 years old.

DETAILED DESCRIPTION:
The BRAIN-M project is driven by the idea that understanding the mechanisms through which muscle and brain interact could offer new approaches to magnifying the beneficial and detrimental effects of exercise training on health at older age. Specifically, the investigators aim at identifying brain, blood, and muscle biomarkers that could serve as predictors of response to exercise training at either cognitive, brain, muscle or physical performance levels and study the associations between biomarkers in order to suggest a physiological model of brain-muscle and muscle-brain crosstalk in ageing. 60 male older adults (60-75y old) will be included in either 12 weeks of high-intense blood-flow restriction training (n = 20), muscle damaging resistance training (n = 20) or no exercise (n = 20). The control group will be asked to maintain their usual lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* healthy male older adults
* able to speak and read fluent Lithuanian
* living in community during the study

Exclusion Criteria:

* cognitive and neurological disorders (e.g. dementia, stroke, Parkinson, multiple sclerosis)
* previous lower extremity injury
* diabetes mellitus type I or II
* no oncologic disease
* no bone fractures in the previous year
* deep vein thrombosis
* cardiovascular disorders (e.g. congestive heart failure, angina pectoris, uncontrolled arrhythmia, history of myocardial infarction or coronary bypass grafting in the past year)
* obesity (BMI >30kg/m²)
* chronic fatigue, chronic headache, or chronic dizziness
* ineligibility to MRI scanning (e.g. due to claustrofobia or metal implants)
* The participants should not be engaged in any regular exercise programme during the previous 6 months (according to IPAQ), but able to perform 10 sit-ups
* Any other consideration that interferes with the study aims and/or risk to the participant, at the discretion of the researcher

Ages: 60 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-10-15 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function on the Switching task (executive function) | Before first exercise bout, immediately after first exercise bout, 1 hour after the first exercise bout and after the 12 week intervention period
  The switching task is a complex task where subjects need to switch (executive function) between a manikin task (visuospatial skill, attention and problem solving) and a mathematical computation task (mathematical computation skill, concentration and working memory).

SECONDARY OUTCOMES:
Change in cognitive function on the 2-Choice Reaction time (processing speed), Go/No-Go (inhibition) or 6 letter Memory Search (memory) test | Before first exercise bout, immediately after first exercise bout, 1 hour after the first exercise bout and after the 12 week intervention period
  Cognitive functioning will be assessed with the Automated Neuropsychological Assessment Metrics 4 (ANAM4) cognitive test battery, testing several cognitive domains.
Changes in lactate levels | Before first exercise bout, immediately after first exercise bout, 1 hour after the first exercise bout
  Capillary lactate levels will be measured in the acute exercise test.
Changes in blood serum levels of TNFalpha and syndecan | Before first exercise bout, immediately after first exercise bout, 1 hour after the first exercise bout
  We will use enzyme-linked immunosorbent assays (ELISAs) to measure acute changes in TNFalpha, and syndecan before and after the first exercise bout.
Changes in blood plasma levels of BDNF | Before first exercise bout, immediately after first exercise bout, 1 hour after the first exercise bout and after the 12 week intervention period
  We will use enzyme-linked immunosorbent assays (ELISAs) to measure acute and chronic changes in BDNF before and after the first exercise bout; and after 12 weeks intervention
Changes in blood serum levels of IGF-1, IL-6 and kynurenine | Before and after the 12 week intervention period
  We will use enzyme-linked immunosorbent assays (ELISAs) to measure chronic changes in IGF-1, IL-6 and kynurenine before and after 12 weeks intervention
Changes in blood CK levels | Before first exercise bout and every 3 weeks for a total of 7 times 48 hours after the eccentric-only training session in the MDRT group.
  Blood CK levels will be measured in the MDRT group 48 hours after each eccentric-only training session to assess the muscle damaging effect/repeated bout effect.
Changes in muscle contractile characteristics (with tensiomyography (TMG)) | Before and after the 12 week intervention period
  Muscle involuntary contractile characteristics of the lower-limb muscles-the rectus femoris (RF), vastus medialis (VM), vastus lateralis (VL), biceps femoris (BF), semitendinosus (ST), tibialis anterior (TA), gastrocnemius medialis (GM) and gastrocnemius lateralis (GL)-will be recorded by measuring the response of these muscles to an induced electric stimulus (provoked by two self-adhesive electrodes) using TMG equipment on both the left and right lower extremities.
Changes in BMI | Before and after the 12 week intervention period
  Weight and height will be combined to report BMI in kg/m^2
Changes in body fat % | Before and after the 12 week intervention period
  body fat % will be measured using bio-impedance analysis (Tanita)
Changes in SMI | Before and after the 12 week intervention period
  Skeletal muscle mass index (SMI, kg/m^2) will be measured using bio-impedance analysis (Tanita)
Changes in fat free mass | Before and after the 12 week intervention period
  Fat free mass (kg) will be measured using bio-impedance analysis (Tanita)
Changes in patellar tendon crossectional area | Before and after the 12 week intervention period
  Ultrasound will be used to assess the crossectional area (cm^2) of the pattella tendon
Changes in patellar tendon stiffness | Before and after the 12 week intervention period
  While producing isometric knee extension force, ultrasound will be used to assess patellar tendon distension, which is a measure of tendon stiffness.
Changes in quadriceps muscle fascicle length | Before and after the 12 week intervention period
  Ultrasound will be used to quantify muscle geometrical properties such as fascicle length (cm).
Changes in quadriceps muscle fascicle angle | Before and after the 12 week intervention period
  Ultrasound will be used to quantify muscle geometrical properties such as fascicle angle (°).
Changes in quadriceps muscle thickness | Before and after the 12 week intervention period
  Ultrasound will be used to quantify muscle geometrical properties such as quadriceps muscle thickness.
Changes in quadriceps muscle cross-sectional area | Before and after the 12 week intervention period
  MRI will be used to measure muscle cross-sectional volume changes of the quadriceps muscles
Changes in quadriceps muscle fiber type | Before and after the 12 week intervention period
  H-MRS (proton magnetic resonance spectroscopy) will be used to measure fiber type in the quadriceps muscle
Changes in quadriceps muscle intramuscular fat | Before and after the 12 week intervention period
  H-MRS (proton magnetic resonance spectroscopy) will be used to measure intramuscular fat in the quadriceps muscle
Changes in brain gray matter volume (with magnetic resonance imaging) | Before and after the 12 week intervention period
  MRI will be used to measure changes in gray matter volume using T1 images
Changes in brain white matter volume (with magnetic resonance imaging) | Before and after the 12 week intervention period
  MRI will be used to measure changes in white matter integrity using DTI sequence
Changes in brain neural integrity (with proton magnetic resonance spectroscopy) | Before and after the 12 week intervention period
  H-MRS will be used to measure changes in N-acetylaspartate levels in specific brain regions: right dorsolateral prefrontal cortex, left hippocampus and left primary sensorimotor cortex.
Changes in brain neuroinflammation (with proton magnetic resonance spectroscopy) | Before and after the 12 week intervention period
  H-MRS will be used to measure changes in myo-inositol levels in specific brain regions: right dorsolateral prefrontal cortex, left hippocampus and left primary sensorimotor cortex.
Changes in brain neuroplasticity marker (with proton magnetic resonance spectroscopy) | Before and after the 12 week intervention period
  H-MRS will be used to measure changes in Glx in specific brain regions: right dorsolateral prefrontal cortex, left hippocampus and left primary sensorimotor cortex.
Changes in balance (with posturography on Kistler platform) | Before and after the 12 week intervention period
  Balance will be assessed in four different positions (two legs stance vs Romberg stance with eyes open vs closed) with or without a cognitive task to measure dual task effects.
Changes in handgrip strength | Before and after the 12 week intervention period
  Handgrip strength will be measured using Jamar dynamometry
Changes in maximal isometric strength (with Biodex) | Before and after the 12 week intervention period
  Knee extension/flexion maximal isometric strength (N) will be measured using Biodex.
Changes in isokinetic peak torque (with Biodex) | Before and after the 12 week intervention period
  Knee extension/flexion isokinetic peak torque measurements will be done at 60°/s
Changes in rate of force development (with Biodex) | Before and after the 12 week intervention period
  Rate of force development will be measured during maximal knee extension/flexion movement.
Changes in physical performance (with the Fitness Fullerton Test battery for the Senior) | Before and after the 12 week intervention period
  Determination of motor control tasks relevant to daily life activities. A selection of tests, including the sit-to-stance test, timed up-and-go test, and other physical tests
Changes in subjective quality of life (patient reported outcome questionnaires) | Before and after the 12 week intervention period
  Quality of life will be assessed using the World Health Organisation 100 (WHO 100) questionnaire
Changes in nutrition (patient reported outcome questionnaires) | Before and after the 12 week intervention period
  We will use a selection of patient reported outcome measures to evaluate their nutrition (using the Actual nutrition registration questionnaire).
Changes in subjective sleep quality (patient reported outcome questionnaires) | Before and after the 12 week intervention period
  We will use a selection of patient reported outcome measures to evaluate their quality of sleep (using the Stanford sleep quality scale).
Changes in reported physical activity levels (patient reported outcome questionnaires) | Before and after the 12 week intervention period
  We will assess physical activity levels using the International Physical Activities Questionnaire (IPAQ)

CONTACTS AND LOCATIONS:
Overall Officials: Nerijus Masiulis, PhD, Principal Investigator — Lithuanian Sports University
Locations (1):
- Lithuanian Sports University, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No